CLINICAL TRIAL: NCT05103527
Title: Dorsal Root Ganglion Stimulation Outcomes for the Treatment of Mechanical Knee Pain Among Patients With Osteoarthritis of the Surgical and Non-surgical Knee
Brief Title: Dorsal Root Ganglion Stimulation for the Treatment of Arthritic Knee Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kenneth B Chapman (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor-Investigator, Kenneth B Chapman, Principle Investigator, Spine and Pain Institute of New York
Organization: Spine and Pain Institute of New York (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRG-S for Knee OA
Record Dates: First submitted 2021-09-23; First posted 2021-11-02 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Knee Osteoarthritis; Knee Pain Chronic; Knee Arthritis; Knee Arthropathy
Keywords: Dorsal Root Ganglion Stimulation; knee pain; knee arthritis; osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Subjects will undergo one week DRG-S trial, and for those that respond as defined by 50% or greater pain relief, proceed to DRG-S permanent device system implant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Non-operated Knee Osteoarthritis (Experimental): DRG-S for knee osteoarthritis patients with no history of knee surgery
  Interventions: Device: Dorsal Root Ganglion Stimulation
- Surgically Repaired Knee Osteoarthritis (Experimental): DRG-S for knee osteoarthritis patients with history of surgical repair of the knee
  Interventions: Device: Dorsal Root Ganglion Stimulation

INTERVENTIONS:
Device: Dorsal Root Ganglion Stimulation — Stimulation at L2, L3, L4 and S1 spinal levels

SUMMARY:
Dorsal root ganglion stimulation (DRG-S) may be able to treat mechanical pain caused by tissue injury or damage such as trauma or arthritis in addition to pain caused by nerve dysfunction or injury. The purpose of this study is to determine if dorsal root ganglion stimulation (DRG-S) can effectively treat arthritic pain of the knee.

DETAILED DESCRIPTION:
Dorsal root ganglion stimulation (DRG-S) is a novel form of neuromodulation used to treat chronic neuropathic pain of the groin and lower extremities related to complex regional pain syndrome type I or II (causalgia). DRG-S has shown promise in treating traditionally mixed neuropathic and mechanical pain syndromes such as axial low back pain, suggesting DRG-S may be able to treat mechanical pain in addition to neuropathic pain. Additionally, in a rodent model of osteoarthritis of the knee, DRG-S alleviated pain related behavior in rats.

This open label feasibility study seeks to evaluate if dorsal root ganglion stimulation with Abbott's Proclaim Dorsal Root Ganglion Neurostimulator System can effectively treat osteoarthritis of the knee. Patients with either osteoarthritis of the non-operated knee or osteoarthritis of the surgically repaired knee will be trialed for one week with dorsal root ganglion stimulation to determine if they positively respond with 50% or greater pain relief. For those patients that have a successful trial, they will be implanted with a permanent stimulation device system and followed for one year post implant to measure knee pain, function and disability, and other related outcomes with sustained DRG-S therapy.

Patients will be seen and evaluated prior to DRG-S trial, and for those that receive permanent implants, re-evaluated at 1, 3, 6, 9 and 12 months after implant.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 21 years old
* Able to provide informed consent
* Primary complaint of chronic knee pain for at least 1 year that interferes with functional activities
* Current pain score on visual analog scale (VAS) intensity ≥60 mm
* One of two groups: 1) Non-operated knee pain patients who want to pursue alternative therapies and delay surgery or are not candidates for knee arthroplasty based on age, frailty, non-operable condition, or poor outcome with other side arthroplasty, or 2) Post traumatic knee pain patients with history of surgical repair (such as meniscal or ligament repair).
* Radiologic confirmation (x-ray/MRI/CT) of Kellgren-Lawrence OA grade of 2 (mild) or 3 (moderate) or 4 (severe) noted within 6 months for the index knee
* Continued pain in the target knee despite at least 3 months of conservative treatments with documented failure of physical therapy and standard conservative therapy, including trials of at least two different classes of analgesic medication
* Failure of one or more prior interventional pain procedures such intraarticular corticosteroid or hyaluronidase knee injections, cooled radiofrequency ablation therapy, or regenerative medicine or prior surgery of the knee

Exclusion Criteria:

* Non-English speaking
* Douleur neuropathique 4 (DN4) score ≥4
* Receiving opioid analgesic medication at a dose of ≥90 mg oral morphine equivalents
* Workers' compensation or no-fault insurance
* Signs or symptoms of active infection in the index knee joint
* Pregnancy
* BMI >45
* Presence of any contraindication for DRG stimulation, including neurological, medical, psychiatric, or social conditions.
* Widespread pain conditions like fibromyalgia
* Autoimmune/Inflammatory arthritic conditions such as Rheumatoid and psoriatic arthritis and other allied disorders (sjogren, felty, inflammatory bowl disease etc)
* Collagen diseases (systemic lupus erythematosus, Scleroderma, etc)
* Infectious arthritis
* Evidence of prespecified joint safety conditions (eg, rapidly progressive OA, subchondral insufficiency fracture, osteonecrosis, pathologic fracture) in the index knee on screening radiographs
* Scheduled for or anticipating any surgery during the trial period

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Treatment success rate at 3 months | 3 months post-implant
  Percent of DRG-S implanted patients that successfully respond to stimulation therapy as defined by >=50% reduction in reported pain score from baseline

SECONDARY OUTCOMES:
VAS pain scores | 1-, 3-, 6-, 9-, and 12 months post-implant
  Patient's pain score using standard 10cm pain scale that represents a continuum between "no pain" and "worst pain."
Western Ontario and McMaster Universities Arthritis Index (WOMAC) for knee pain patients | 1-, 3-, 6-, 9-, and 12 months post-implant
  At each study visit, subjects will complete WOMAC survey which assesses pain, stiffness, and function in patients with OA of the knee.
European Quality of Life 5 Dimension (EQ-5D) | 1-, 3-, 6-, 9-, and 12 months post-implant
  At each study visit, subjects will complete EQ-5D survey which assesses health-related quality of life
Short Form 36 Mental Component Summary (SF-36 MCS) | 1-, 3-, 6-, 9-, and 12 months post-implant
  At each study visit, subjects will complete SF-36 MCS survey which assesses mental health
Pain Disability Index (PDI) | 1-, 3-, 6-, 9-, and 12 months post-implant
  At each study visit, subjects will complete PDI survey which assesses pain-related disability
Patient Global Impression of Change (PGIC) | 1-, 3-, 6-, 9-, and 12 months post-implant
  At each study visit, subjects will complete PDI survey which assesses patient's belief about the efficacy of treatment
Medication Dosage | 1-, 3-, 6-, 9-, and 12 months post-implant
  Patient's dose of narcotic analgesics measured in morphine milligram equivalents (MME) and non-narcotic analgesics and dosages
Timed Up and Go (TUG) | 1-, 3-, 6-, 9-, and 12 months post-implant
  Video recordings of motor task exams will be used to measure TUG, a performance-based measure of functional mobility which measures the time for subject to rise from a chair, walk three meters, turn around, return to the chair, and sit down.
Knee Range of Motion (ROM) | 1-, 3-, 6-, 9-, and 12 months post-implant
  Video recordings of motor task exams will be used to measure ROM of the index knee
Serum concentrations of molecular biomarkers | 3-, 6-, and 12-months post-implant
  Serum concentrations of molecular biomarkers related to knee OA including but not limited to C-telopeptide of crosslinked collagen type I and type II (CTX-I and CTX-II)
Kellgren-Lawrence System for Classification of Osteoarthritis | 6- and 12-months post-implant
  Radiologic classification of subject's knee x-ray to grade progression/severity of osteoarthritis
Treatment success rate at other post-implant timepoints | 1-, 6-, 9-, and 12-months post-implant
  Percent of DRG-S implanted patients that successfully respond to stimulation therapy as defined by >=50% reduction in reported pain score from baseline

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 12 months post-implant
  All complications of DRG-S trial, implant, and stimulation therapy will be reported

CONTACTS AND LOCATIONS:
Locations (1):
- The Spine and Pain Institute of New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu G, Segel I, Zhang Z, Hogan QH, Pan B. Dorsal Root Ganglion Stimulation Alleviates Pain-related Behaviors in Rats with Nerve Injury and Osteoarthritis. Anesthesiology. 2020 Aug;133(2):408-425. doi: 10.1097/ALN.0000000000003348. PMID 32433276
- [Background] Bjerre-Bastos JJ, Bay-Jensen A-C, Karsdal MA, Byrjalsen I, Andersen JR, Riis BJ, et al. Biomarkers of bone and cartilage turnover CTX-I and CTX-II predict total joint replacements in osteoarthritis. Osteoarthr Cartil [Internet]. 2019;27(2019):S31-2. Available from: https://doi.org/10.1016/j.joca.2019.02.046
- [Background] Convill JG, Tawy GF, Freemont AJ, Biant LC. Clinically Relevant Molecular Biomarkers for Use in Human Knee Osteoarthritis: A Systematic Review. Cartilage. 2021 Dec;13(1_suppl):1511S-1531S. doi: 10.1177/1947603520941239. Epub 2020 Jul 17. PMID 32680434
- [Background] Adhikary SD, Liu WM, Memtsoudis SG, Davis CM 3rd, Liu J. Body Mass Index More Than 45 kg/m(2) as a Cutoff Point Is Associated With Dramatically Increased Postoperative Complications in Total Knee Arthroplasty and Total Hip Arthroplasty. J Arthroplasty. 2016 Apr;31(4):749-53. doi: 10.1016/j.arth.2015.10.042. Epub 2015 Nov 10. PMID 26652477
- [Background] van Bussel CM, Stronks DL, Huygen FJPM. Dorsal Column Stimulation vs. Dorsal Root Ganglion Stimulation for Complex Regional Pain Syndrome Confined to the Knee: Patients' Preference Following the Trial Period. Pain Pract. 2018 Jan;18(1):87-93. doi: 10.1111/papr.12573. Epub 2017 May 4. PMID 28334499
- [Background] Kallewaard JW, Edelbroek C, Terheggen M, Raza A, Geurts JW. A Prospective Study of Dorsal Root Ganglion Stimulation for Non-Operated Discogenic Low Back Pain. Neuromodulation. 2020 Feb;23(2):196-202. doi: 10.1111/ner.12937. Epub 2019 Mar 1. PMID 30821901
- [Background] Huygen F, Liem L, Cusack W, Kramer J. Stimulation of the L2-L3 Dorsal Root Ganglia Induces Effective Pain Relief in the Low Back. Pain Pract. 2018 Feb;18(2):205-213. doi: 10.1111/papr.12591. Epub 2017 Dec 6. PMID 28486758